CLINICAL TRIAL: NCT00819247
Title: A Six Month, Multi-centre, Open-labelled, 1:1:1 Randomised, Parallel Group Study Investigating the Efficacy and Safety of Three Dose Regimens of FE 200486 in Prostate Cancer Patients
Brief Title: The Efficacy and Safety of FE 200486 in Treatment of Patients Suffering From Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Clinical Development Support, Ferring Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FE200486 CS02
Record Dates: First submitted 2009-01-07; First posted 2009-01-08 (Estimated); Results first posted 2009-03-31 (Estimated); Last update posted 2023-11-09 (Actual); Status verified 2011-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Degarelix 80/80 + 40 (Experimental): Loading doses of Degarelix 80 mg (20 mg/mL) on Days 0 and 3. Maintenance doses of 40 mg (20 mg/mL) given on days 28, 56, 84, 112 and 140.
  Interventions: Drug: Degarelix
- Degarelix 40/40 + 40 (Experimental): Loading doses of Degarelix 40 mg (20 mg/mL) on Days 0 and 3. Maintenance doses of 40 mg (20 mg/mL) given on days 28, 56, 84, 112 and 140.
  Interventions: Drug: Degarelix
- Degarelix 80 + 20 (Experimental): Loading dose of Degarelix 80 mg (20 mg/mL) on Day 0. Maintenance doses of 20 mg (10 mg/mL) given on days 28, 56, 84, 112 and 140.
  Interventions: Drug: Degarelix

INTERVENTIONS:
Drug: Degarelix — Given as a subcutaneous injection.
  Other Names: FE 200486

SUMMARY:
The purpose of this trial was to select a dose of degarelix (FE 200486). Three groups of patients were treated for six months on different doses. The patients had blood samples taken and measured for Testosterone in order to determine the most efficient dose to provide fast and sustained castration. The patients came to the clinic for 16 visits and dependent on the blood sample results they were invited to return for additional blood samples on a two weekly basis.

DETAILED DESCRIPTION:
Degarelix was not FDA regulated at the time of the trial. After completion of the trial degarelix has been approved by the FDA and is thus an FDA regulated intervention.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent before any trial related activity
* Proven prostate cancer with a need for endocrine treatment
* Testosterone level within the normal range for the age

Exclusion Criteria:

* Previous or current hormonal treatment of prostate cancer
* Candidate for prostatectomy or radiotherapy
* History of severe asthma, anaphylactic reactions or Quincke's Oedema
* Hypersensitivity towards any component of FE200486
* Cancer disease within the last ten years except for prostate cancer and some skin cancers
* Presenting with significant neurological, gastrointestinal, renal, hepatic, cardiovascular, psychological, pulmonary, metabolic, endocrine, haematological, dermatological or infectious disorder. In addition any other condition such as excessive alcohol or drug abuse that may interfere with trial participation or influence the conclusion of the trial as judged by the investigator
* Mental incapacity or language barrier
* Having received an investigational product within the last 12 weeks preceding the trial
* Previous participation in this trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2001-03; Primary Completion 2002-05 (Actual); Study Completion 2002-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (16):
- United Kingdom (16):
  - Ayr Hospital, Ayr
  - Bristol Royal Infirmary, Bristol
  - Southmead Hospital, Bristol
  - St. Richards Hospital, Chichester
  - Glan Clwyd Hospital, Denbighshire
  - Ninewells Hospital, Dundee
  - Southern General Hospital, Glasgow
  - Leicester General Hospital, Leicester
  - Chelsea and Westminster Hospital, London
  - Kings College Hospital, London
  - St. Bartholemews Hospital, London
  - Derriford Hospital, Plymouth
  - Lister Hospital, Stevenage
  - Stirling Royal Infirmary, Stirling
  - Morriston Hospital, Swansea
  - Pindersfields General Hospital, Wakefield

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One hundred and fifty-nine participants were screened. One hundred and twenty-nine participants were randomised, two of these participants withdrew before receiving any treatment.
Groups:
- Degarelix 80/80 + 40: Loading doses of Degarelix 80 mg on Days 0 and 3. Maintenance doses of 40 mg given on days 28, 56, 84, 112 and 140.
- Degarelix 40/40 + 40: Loading doses of Degarelix 40 mg on Days 0 and 3. Maintenance doses of 40 mg given on days 28, 56, 84, 112 and 140.
- Degarelix 80 + 20: Loading dose of Degarelix 80 mg on Day 0. Maintenance doses of 20 mg given on days 28, 56, 84, 112 and 140.
Period: Overall Study
Arm/Group | Degarelix 80/80 + 40 | Degarelix 40/40 + 40 | Degarelix 80 + 20
Started | 43 | 46 | 40
Randomized | 43 | 46 | 40
Intent-to-treat Population | 42 (One randomised participant withdrew at Day 1.) | 46 | 39 (One randomised participant withdrew at Day 1.)
Per Protocol Population | 38 (One participant- baseline testosterone outside normal range. Three participants- prohibited drugs.) | 44 (Two participants - prohibited drugs) | 38 (One participant - baseline testosterone outside normal range.)
Completed | 32 | 30 | 26
Not Completed | 11 | 16 | 14
Not completed — Adverse Event | 0 | 5 | 3
Not completed — Insufficient testosterone response | 5 | 8 | 10
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 1
Not completed — Mistakenly withdrawn | 0 | 1 | 0
Not completed — Bad prostate-specific antigen response | 3 | 2 | 0
Not completed — Other | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Degarelix 80/80 + 40 | Degarelix 40/40 + 40 | Degarelix 80 + 20 | Total
Number analyzed (Participants) | 43 | 46 | 40 | 129
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 7 | 18
  >=65 years | 37 | 41 | 33 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.4 (6.6) | 73.7 (7.2) | 71.8 (7.1) | 72.7 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 43 | 46 | 40 | 129
Race/Ethnicity, Customized [Number; unit: participants]
  White | 42 | 43 | 37 | 122
  Black | 1 | 3 | 1 | 5
  Oriental / Asian | 0 | 0 | 0 | 0
  Afro-carribean | 0 | 0 | 1 | 1
  Indian | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United Kingdom | 43 | 46 | 40 | 129
Participant Counts by Gleason Score [Number; unit: participants] — The Gleason score is a system of grading the aggressiveness of the prostate cancer and how fast it is likely to grow and spread. Scale is 2-10, with low numbers being the least aggressive and 10 being the most aggressive.
  participants
    unknown | 1 | 1 | 1 | 3
    2-4 | 3 | 4 | 2 | 9
    5-6 | 11 | 7 | 11 | 29
    7-10 | 28 | 34 | 26 | 88
Stage of Prostate Cancer [Number; unit: participants] — Prostate cancer stage was classified to describe the extent of cancer. Localized refers to tumors without involvement of lymph nodes or metastasis. Advanced localized can be larger tumors that may involve the lymph nodes but no metastasis. Metastatic are more advanced cancers that are spreading beyond the original tumor.
  participants
    Localized | 8 | 9 | 5 | 22
    Locally advanced | 21 | 21 | 18 | 60
    Metastatic | 11 | 14 | 17 | 42
    Not classifiable | 3 | 2 | 0 | 5
Body Mass Index [Median (Full Range); unit: kilogram per square meter] — Body mass index is a measure of body fat based on height and weight
  kilogram per square meter | 26.2 [18.0 to 36.4] | 26.6 [17.4 to 40.9] | 25.2 [19.8 to 34.1] | 26.1 [17.4 to 40.9]
Days Since Diagnosis of Prostate Cancer [Mean (Standard Deviation); unit: days] — The number of days passed since a diagnosis of prostate cancer was made for each participant.
  days | 52.7 (116.0) | 153.8 (518.1) | 88.8 (370.0) | 99.9 (377.2)
Serum Prostate-Specific Antigen level [Median (Full Range); unit: nanogram/milliliter] — Prostate-specific antigen (PSA) is a protein produced by the cells of the prostate gland. The PSA test measures the level of PSA in the blood. High PSA levels have a positive correlation to prostate cancer.
  nanogram/milliliter | 50.3 [23.2 to 2580] | 64.6 [18.1 to 2380] | 82.9 [23.7 to 12500] | 61.1 [18.1 to 12500]
Serum Testosterone level [Median (Full Range); unit: nanogram/milliliter] — Testosterone is a steroid hormone from the androgen group, and the principal male sex hormone. This test measures the amount of testosterone in the blood. Androgen deprivation is used to manage prostate cancer.
  nanogram/milliliter | 3.7 [2.13 to 7.63] | 4.1 [1.21 to 7.84] | 4.8 [1.58 to 8.94] | 4.0 [1.21 to 8.94]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Testosterone <0.5 Nanogram/Milliliter
Time Frame: Weeks 1,2,4,8,12,16,20,24
Population: Per protocol population
Measure: Number; unit: participants
Arm/Group | Degarelix 80/80 + 40 | Degarelix 40/40 + 40 | Degarelix 80 + 20
Number analyzed (Participants) | 38 | 44 | 38
participants
  Week 1 (n=38, 44, 38) | 38 | 32 | 27
  Week 2 (n=38, 44, 38) | 38 | 36 | 33
  Week 4 (n=38, 36, 33) | 38 | 35 | 31
  Week 8 (n=36, 36, 31) | 36 | 36 | 31
  Week 12 (n=34, 34, 31) | 34 | 34 | 30
  Week 16 (n=34, 32, 30) | 33 | 31 | 27
  Week 20 (n=33, 31, 28) | 31 | 30 | 25
  Week 24 (n=31, 29, 25) | 28 | 27 | 22

2. Secondary Outcome: Number of Participants With Testosterone < 0.5 Nanogram/Milliliter at All Visits Between Weeks 4-24
Time Frame: Weeks 4-24
Population: Per protocol population
Measure: Number; unit: participants
Arm/Group | Degarelix 80/80 + 40 | Degarelix 40/40 + 40 | Degarelix 80 + 20
Number analyzed (Participants) | 32 | 29 | 27
participants | 28 | 27 | 20

3. Secondary Outcome: Number of Participants Not Meeting a Testosterone Withdrawal Criterion Between Weeks 4-24
Description: Participants with one testoterone value > 1.0 nanogram/millliliter or two consecutive values between 0.5-1.0 nanogram/milliliter were withdrawn from the study due to insufficient response.
Time Frame: Weeks 4-24
Population: Per protocol population
Measure: Number; unit: participants
Arm/Group | Degarelix 80/80 + 40 | Degarelix 40/40 + 40 | Degarelix 80 + 20
Number analyzed (Participants) | 32 | 29 | 27
participants | 29 | 29 | 25

4. Secondary Outcome: Number of Participants Who Met the Withdrawl Criteria for Prostate-specific Antigen
Description: Participants who met at least one of the three criteria for inadequate response on prostate-specific antigen levels (PA). (1) >=25 percent and/or 50 nanogram/milliliter compared to baseline (2) reduction of <=50% compared to baseline at week 12 (3) increase of >=10 nanogram/milliliter compared to nadir from week 4.
Time Frame: Six months
Population: per protocol population
Measure: Number; unit: participants
Arm/Group | Degarelix 80/80 + 40 | Degarelix 40/40 + 40 | Degarelix 80 + 20
Number analyzed (Participants) | 38 | 44 | 38
participants
  >=25% and/or 50 ng/mL compared to baseline | 0 | 0 | 0
  <=50% compared to baseline | 0 | 0 | 0
  >=10 ng/mL compared to nadir | 1 | 6 | 1

5. Secondary Outcome: Number of Participants With Normal Prostate-specific Antigen Levels During the Study
Description: The number of participants whose prostate-specific antigen levels at weeks 12 and 24 were <= 4 nanogram/millliliter (normal level).
Time Frame: Weeks 12, 24
Population: Per Protocol Population
Measure: Number; unit: participants
Arm/Group | Degarelix 80/80 + 40 | Degarelix 40/40 + 40 | Degarelix 80 + 20
Number analyzed (Participants) | 38 | 44 | 38
participants
  Week 12 (n=34, 34, 31) | 18 | 18 | 16
  Week 24 (n=31, 29, 25) | 18 | 18 | 17

6. Secondary Outcome: The Number of Participants With Abnormal Liver Function Tests
Description: The number of participants who had abnormal [defined as above upper limit of normal range (ULN)] alanine aminotransferase (ALT), participants with ALT increases > 3x ULN, and participants with ALT increases > 3x ULN with concurrent increases in bilirubin > 1.5 ULN.
Time Frame: Six months
Population: Randomized (Safety) population
Measure: Number; unit: participants
Arm/Group | Degarelix 80/80 + 40 | Degarelix 40/40 + 40 | Degarelix 80 + 20
Number analyzed (Participants) | 43 | 46 | 40
participants
  Alanine aminotransferase (ALT) above upper limit | 13 | 14 | 12
  ALT levels >3x upper limit | 0 | 1 | 1
  ALT levels >3x and bilirubin >1.5x upper limit | 0 | 0 | 1

7. Secondary Outcome: Percentage Change in Vital Signs and Body Weight
Description: Percentage changes in vital signs (systolic and diastolic blood pressure and pulse) and body weight at the end of trial as compared to baseline.
Time Frame: Baseline and Six months
Population: Safety population.
Measure: Median (Full Range); unit: percentage
Arm/Group | Degarelix 80/80 + 40 | Degarelix 40/40 + 40 | Degarelix 80 + 20
Number analyzed (Participants) | 43 | 46 | 40
percentage
  Diastolic blood pressure | 0.0 [-24 to 43] | -0.6 [-45 to 55] | 0.0 [-38 to 32]
  Systolic blood pressure | -3.7 [-19 to 23] | -2.4 [-25 to 57] | 0.0 [-39 to 29]
  Pulse | -3.1 [-26 to 42] | 0.0 [-23 to 30] | -1.5 [-29 to 44]
  Weight | 2.8 [-11 to 24] | 2.6 [-7 to 17] | 3.5 [-23 to 17]

ADVERSE EVENTS:
Arm/Group | Degarelix 80/80 + 40 | Degarelix 40/40 + 40 | Degarelix 80 + 20
Serious Adverse Events (participants affected / at risk) | 3 | 8 | 6
Other Adverse Events (participants affected / at risk) | 38 | 38 | 32
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Degarelix 80/80 + 40 | Degarelix 40/40 + 40 | Degarelix 80 + 20
Anaemia (Blood and lymphatic system disorders) | 1/43 (1) | 1/46 (1) | 0/40 (0)
Angina pectoris (Cardiac disorders) | 1/43 (1) | 0/46 (0) | 1/40 (1)
Myocardial infarction (Cardiac disorders) | 1/43 (1) | 1/46 (1) | 0/40 (0)
Cardiac failure congestive (Cardiac disorders) | 1/43 (1) | 0/46 (0) | 0/40 (0)
Nausea (Gastrointestinal disorders) | 0/43 (0) | 1/46 (2) | 0/40 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0/43 (0) | 1/46 (1) | 0/40 (0)
Vomiting (Gastrointestinal disorders) | 0/43 (0) | 1/46 (1) | 0/40 (0)
Asthenia (General disorders) | 0/43 (0) | 1/46 (1) | 0/40 (0)
Catheter related complication (General disorders) | 0/43 (0) | 1/46 (1) | 0/40 (0)
Condition aggravated (General disorders) | 0/43 (0) | 0/46 (0) | 1/40 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0/43 (0) | 0/46 (0) | 1/40 (1)
Hypersensitivity (Immune system disorders) | 0/43 (0) | 1/46 (1) | 0/40 (0)
Lobar pneumonia (Infections and infestations) | 0/43 (0) | 1/46 (1) | 0/40 (0)
Sepsis (Infections and infestations) | 0/43 (0) | 1/46 (1) | 0/40 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0/43 (0) | 1/46 (1) | 0/40 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0/43 (0) | 0/46 (0) | 1/40 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/43 (0) | 1/46 (1) | 0/40 (0)
Cerebral haemorrhage (Nervous system disorders) | 0/43 (0) | 1/46 (1) | 0/40 (0)
Cerebrovascular accident (Nervous system disorders) | 0/43 (0) | 0/46 (0) | 1/40 (1)
Syncope (Nervous system disorders) | 0/43 (0) | 1/46 (1) | 0/40 (0)
Depression (Psychiatric disorders) | 1/43 (1) | 0/46 (0) | 1/40 (1)
Alcoholism (Psychiatric disorders) | 1/43 (1) | 0/46 (0) | 0/40 (0)
Bladder obstruction (Renal and urinary disorders) | 0/43 (0) | 0/46 (0) | 1/40 (1)
Calculus bladder (Renal and urinary disorders) | 0/43 (0) | 1/46 (1) | 0/40 (0)
Dysuria (Renal and urinary disorders) | 0/43 (0) | 0/46 (0) | 1/40 (1)
Urine flow decreased (Renal and urinary disorders) | 0/43 (0) | 1/46 (1) | 0/40 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0/43 (0) | 1/46 (2) | 0/40 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Degarelix 80/80 + 40 | Degarelix 40/40 + 40 | Degarelix 80 + 20
Diarrhoea (Gastrointestinal disorders) | 6/43 (9) | 2/46 (2) | 2/40 (4)
Constipation (Gastrointestinal disorders) | 3/43 (3) | 1/46 (1) | 1/40 (1)
Inguinal hernia (Gastrointestinal disorders) | 1/43 (1) | 1/46 (1) | 2/40 (2)
Dyspepsia (Gastrointestinal disorders) | 0/43 (0) | 1/46 (1) | 2/40 (2)
Abdominal pain (Gastrointestinal disorders) | 0/43 (0) | 0/46 (0) | 2/40 (2)
Fatigue (General disorders) | 2/43 (2) | 4/46 (5) | 0/40 (0)
Suprapubic pain (General disorders) | 0/43 (0) | 0/46 (0) | 2/40 (2)
Nasopharyngitis (Infections and infestations) | 5/43 (6) | 7/46 (7) | 5/40 (5)
Urinary tract infection (Infections and infestations) | 3/43 (5) | 1/46 (1) | 2/40 (2)
Weight increased (Investigations) | 0/43 (0) | 0/46 (0) | 2/40 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3/43 (3) | 3/46 (3) | 2/40 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0/43 (0) | 3/46 (3) | 0/40 (0)
Headache (Nervous system disorders) | 4/43 (5) | 2/46 (2) | 3/40 (4)
Lethargy (Nervous system disorders) | 2/43 (2) | 3/46 (4) | 1/40 (1)
Dysuria (Renal and urinary disorders) | 3/43 (4) | 0/46 (0) | 2/40 (4)
Pollakiuria (Renal and urinary disorders) | 0/43 (0) | 1/46 (1) | 2/40 (2)
Testicular atrophy (Reproductive system and breast disorders) | 3/43 (3) | 2/46 (2) | 4/40 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 2/43 (2) | 2/46 (2) | 2/40 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3/43 (3) | 3/46 (3) | 1/40 (1)
Skin reaction (Skin and subcutaneous tissue disorders) | 3/43 (3) | 0/46 (0) | 0/40 (0)
Hot flush (Vascular disorders) | 21/43 (22) | 21/46 (21) | 22/40 (25)
Flushing (Vascular disorders) | 4/43 (4) | 6/46 (6) | 2/40 (2)
Hypertension (Vascular disorders) | 3/43 (3) | 2/46 (2) | 1/40 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript.